CLINICAL TRIAL: NCT02284438
Title: Innovation Against Infection - Device Related Infections - Part ETT
Brief Title: Biofilm Formation on Different Endotracheal Tube Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Vinnova (Other Government); Bactiguard AB (Industry)
Responsible Party: Principal Investigator, Bengt Klarin, MD Consultant, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IMI-ETT
Record Dates: First submitted 2014-10-21; First posted 2014-11-06 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Insufficiency; Ventilator-associated Pneumonia
Keywords: ETT; Biofilm; Mechanical ventilation; Critical illness; Ventilator-associated pneumonia
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Ventilator-Associated; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biofilm formation on ETT (Other): Three different endotracheal tubes uses on intubated mechanical ventilated patients will after extubation be examined regarding biofilm, structure and presence of microbes on the ETTs The different tubes will be used during consecutive time periods The study does not include any interventions concerning the treatment of these critically ill patients
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Endotracheal tube — Three endotracheal tubes with different surfaces will be used

SUMMARY:
Three endotracheal tubes (ETTs) with different surfaces properties will be studied regarding formation and structure of the biofilm formed on those ETTs.

Cultures from oropharynx and tracheal secretions as well as pieces of the ETT will be examined.

Findings from electron microscopy (EM) and microbiology will be analyzed and compared in respect to the three materials.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is a frequent and costly complication to mechanical ventilation in critically ill patients. Aspiration of oropharyngeal secretions and fragments of biofilm from the endotracheal tube are the main causes of VAP.

It is well known that biofilm is formed on medical devices and several initiatives to reduce the development of such biofilms have been taken. However it is still a large clinical problem and colleagues have performed studies to find out the structure of the biofilms formed on the ETT and to what extent microbiological findings correlate to images from EM.

In this study the investigators will compare microbiology and EM images in that same manner.

Three different ETTs will be examined. The investigators will be using each of the three ETTs for a period of time sufficient to retrieve samples from at least 20 ETTs of each kind.

Only one kind of ETT will be used during the specified time period, no randomization. The test will be performed in the order mentioned below A - B - C All of the three tubes are CE-marked (Conformité Européenne) and are available on the market.

ICU patients needing mechanical ventilation will be intubated with the three different devices with different surfaces characteristics.

The tubes are: A - standard Poly vinyl chloride (PVC) tube; B - PVC with a silicon coating; C - PVC with a special metal film coating

ELIGIBILITY:
Inclusion Criteria:

* Patients needing invasive mechanical ventilation through an endotracheal tube

Exclusion Criteria:

* Anticipated need for mechanical ventilation less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Structure, thickness, and presence of microbes of biofilm developed on endotracheal tube | After finished mechanical ventilation and extubation; expected average time on mechanical ventilation 5 days
  Pieces of the tubes examined with electron microscopy and assessed for microbes

SECONDARY OUTCOMES:
White Blood Cell count | From admission to extubation. Expected average 5 days
  Blood samples taken daily
C reactive protein | From admission to extubation. Expected average 5 days
  Blood samples taken daily
Length of stay, ICU and Hospital | Three months from study inclusion
  Length of stay in Hospital and for the ICU stay
Survival | Three months from study inclusion
  For participating patients the status of survival or non survival at days 28 and 90 (three months)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Klarin, MD, PhD, Principal Investigator — Dept Anaesthesiology and Intensive care, Skåne University Hospital, Lund Sweden
Locations (1):
- Intensive Care Unit, Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Results will be published as an article in a scientific journal

REFERENCES:
- [Background] Gil-Perotin S, Ramirez P, Marti V, Sahuquillo JM, Gonzalez E, Calleja I, Menendez R, Bonastre J. Implications of endotracheal tube biofilm in ventilator-associated pneumonia response: a state of concept. Crit Care. 2012 May 23;16(3):R93. doi: 10.1186/cc11357. PMID 22621676
- [Derived] Thorarinsdottir HR, Kander T, Holmberg A, Petronis S, Klarin B. Biofilm formation on three different endotracheal tubes: a prospective clinical trial. Crit Care. 2020 Jun 29;24(1):382. doi: 10.1186/s13054-020-03092-1. PMID 32600373
- See also: Sweden's innovation agency — http://www.vinnova.se/en/
- See also: (Statens Provningsanstalt) SP Technical Research Institute of Sweden, — http://www.sp.se/en/Sidor/default.aspx